CLINICAL TRIAL: NCT00433745
Title: Wilm's Tumor 1 (WT1) Peptide Vaccination for Patients With High Risk Hematological Malignancies
Brief Title: Wilm's Tumor 1 (WT1) Peptide Vaccine for High Risk Hematologic Malignancy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Minoo Battiwalla, M.D., Principal Investigator, National Heart, Lung, and Blood Institute (NHLBI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 070091; 07-H-0091 (Other: National Heart Lung and Blood Institute); NCT00458965 (obsolete NCT alias)
Record Dates: First submitted 2007-02-09; First posted 2007-02-12 (Estimated); Results first posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-06

CONDITIONS: Myelodysplastic Syndrome; Acute Myeloid Leukemia (AML); Chronic Myeloid Leukemia (CML)
Keywords: Myelodysplastic Syndrome (MDS); Acute Myelogenous Leukemia (AML); Chronic Myelogenous Leukemia (CML); Acute Lymphoblastic Leukemia (ALL); Wilm's Tumor-1 Peptide; Leukemia; Myelodysplastic Syndrome; MDS; Acute Myelogenous Leukemia; AML; Chronic Myelogenous Leukemia; CML; Acute Lymphoblastic Leukemia; ALL
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- WT1 Peptide Vaccine (Experimental): WT1 vaccination (9 doses of WT-1:126-134 peptide (in Montanide adjuvant) administered concomitantly with GM-CSF (Sargramostim)
  Interventions: Drug: WT1 Peptide Vaccine

INTERVENTIONS:
Drug: WT1 Peptide Vaccine — WT1 vaccination (9 doses of WT-1:126-134 peptide (in Montanide adjuvant) administered concomitantly with GM-CSF (Sargramostim)
  Other Names: Wilm's tumor 1 vaccine

SUMMARY:
This study will determine the safety and effectiveness of an experimental vaccine in controlling the abnormal growth of cells in patients with myelodysplastic syndrome (MDS, also known as myelodysplasia), acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL), and chronic myeloid leukemia (CML). It will test whether the vaccine can increase the number of immune cells responding to the cancer and thereby slow progression of the illness, improve blood counts, reduce the need for transfusions of blood and platelets, or even achieve a disease remission. The vaccine contains part of a protein that is produced in large amounts by cells of patients with these cancers and an added substance called Montanide that helps the immune system respond to the vaccine. Sargramostim, another substances that boosts the immune response, is also given.

Patients 18 to 85 years of age with MDS, AML, ALL or CML may be eligible for this study. Candidates are screened with a medical history, physical examination, blood tests, chest x-ray and bone marrow biopsy. Women of childbearing age also have a pregnancy test.

Participants undergo the following:

* Chemotherapy entering the study.
* Leukapheresis to collect large amounts of white blood cells for infusion before vaccine administration.
* Participants may need placement of a central line (plastic tube, or catheter) in the upper part of the chest to be used for giving chemotherapy, blood or platelet transfusions, antibiotics and white blood cells, and for collecting blood samples.
* Weekly vaccine injections for nine weeks, given in the upper arm, upper leg or abdomen.
* Sargramostim injections following each vaccination.
* Standard of care treatment for MDS, AML, ALL or CML, which may include blood or platelet transfusions, growth factors, and drugs to control underlying disease and potential side effects of the vaccine.
* Weekly safety monitoring, including vital signs check, brief health assessment, blood tests and observation after the vaccination, on the day of each vaccination.
* Follow-up evaluations with blood tests and chest x-ray 3 weeks after the last vaccine dose and with blood tests and bone marrow biopsy 7 weeks after the last vaccine dose.

DETAILED DESCRIPTION:
Leukemias and the related disorders myelodysplastic syndrome and myeloproliferative diseases represent a wide group of bone marrow stem cell malignancies. Some patients can be cured with chemotherapy or by allogeneic stem cell transplantation. However, standard treatment approaches are not effective for patients who become refractory to chemotherapy, those who relapse after transplantation and those with progressive disease. The management of such patients remains unsatisfactory and requires new treatment approaches other than chemotherapy.

The immunological graft-versus-leukemia (GVL) effect seen after allogeneic stem cell transplantation suggests that stimulating the patient's own T cell responses to hematological malignancies might also retard disease progression and even achieve disease remissions. Wilm's Tumor 1 (WT1) was identified as a target vaccine antigen because this antigen is over-expressed by cluster of differentiation 34 (CD34) plus stem cells of most patients with myeloid and lymphoid malignancies but not by normal marrow cells. A human leukocyte antigen (HLA-A0201) restricted peptide derived from the Wilm's Tumor (WT) protein is anticipated to induce T cell response against MDS and leukemic cells while sparing normal cells. Of note, about 40% of the population is HLA-A0201 positive.

Therefore we propose this Phase II trial, the second in a series of planned peptide vaccine research, which will evaluate the safety associated with an immunotherapy approach of lymphodepletion, lymphocyte infusion, and WT1 vaccination in select patients diagnosed with MDS, AML, ALL and CML. The WT1 vaccination will comprise of 9 doses of WT-1 peptide vaccines (in Montanide adjuvant) administered concomitantly with granulocyte macrophage- colony stimulating factor (GM-CSF) (Sargramostim).

The primary objectives will be to evaluate the efficacy and toxicity associated with the immunotherapy approach of lymphodepletion, lymphocyte infusion, and WT1 vaccination in selected patients with hematological malignancies.

Secondary objectives will include evaluation of disease response by following the numbers of WT1 expressing cells in blood, hematological measurements (reduction in marrow blast cells, changes in blood counts), transfusion dependence, and time to disease progression and survival.

The primary endpoint will be the side effects of treatment (toxicity and number of circulating WT1 specific T cells (efficacy ) measured through week 16 of the study (7 weeks after the last dose of vaccine).

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Diagnosed with

     refractory anemia with excess of blasts (MDS-RAEB).

     or

     refractory anemia with excess of blasts in transformation (MDS-RAEBt).

     or

     secondary acute myelogenous leukemia (AML).

     or

     relapsed or refractory acute or chronic myelogenous leukemias (AML).

     or

     relapsed or refractory chronic myelogenous leukemias (CML) with accelerated phase or blast crisis

     or

     relapsed or refractory acute lymphoblastic leukemia (high risk ALL).

     or

     acute lymphoblastic leukemia (ALL) in complete remission.

     or

     chronic myelomonocytic leukemia (CMML).
  2. Unsuitable for stem cell transplantation (age over sixty or unavailability of a fully-matched donor).

     or

     made an informed decision not to undergo the transplant procedure.

     or

     relapsed AML, CML, MDS or ALL post stem cell transplantation (SCT).
  3. HLA-A0201 positive.
  4. Ages 18 - 85 years.
  5. Off all lympho-ablative chemotherapeutic agents.
  6. All subjects (men and women) must agree to practice abstinence or effective contraception during the study period.

Inclusion Criteria Donor (for post transplant subjects without available donor lymphocyte infusion (DLI) cells):

1. Related donor, HLA identical (6/6) with recipient.
2. Age greater than or equal to 18 or less than or equal to 80 years old.
3. Ability to comprehend the investigational nature of the study and provide informed consent.

EXCLUSION CRITERIA:

1. HIV positive (HIV-infected patients are immune-compromised and it is unlikely that these patients will be capable of mounting an immune response to the vaccine).
2. Treatment with systemic corticosteroids within 7 days prior to study entry.
3. Low bone marrow reserves (less than 20 percent cellularity).
4. Serum creatinine greater than 2.5mg/dl or serum bilirubin greater than 4mg/dl (patients receiving fludarabine).
5. Co-morbidity of such severity that it would preclude the patient's ability to tolerate protocol therapy.
6. Predicted survival less than 3 months.
7. Previous allergic reaction to Montanide Adjuvant.
8. Pregnant or breast feeding (Pregnant and breast-feeding women are excluded from study because the effects of vaccination are not known and may pose a risk to the developing fetus. All female patients will have a urine pregnancy test, and only those that test negative will be allowed on study).
9. Enrolled in another vaccine clinical trial during the study period.
10. Inability to comprehend the investigational nature of the study and provide informed consent.

Exclusion Criteria-Donor (any of the following):

1. Pregnant or lactating.
2. Unfit to receive filgrastim (G-CSF) and undergo apheresis (abnormal blood counts, history of stroke, uncontrolled hypertension).
3. HIV positive.
4. Severe psychiatric illness. Mental deficiency sufficiently severe as to make compliance with the bone marrow transplant (BMT) treatment unlikely and making informed consent impossible.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-02; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Barrett, MD, Principal Investigator — National Institutes of Health- NHLBI
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Rezvani K, Yong AS, Mielke S, Savani BN, Musse L, Superata J, Jafarpour B, Boss C, Barrett AJ. Leukemia-associated antigen-specific T-cell responses following combined PR1 and WT1 peptide vaccination in patients with myeloid malignancies. Blood. 2008 Jan 1;111(1):236-42. doi: 10.1182/blood-2007-08-108241. Epub 2007 Sep 17. PMID 17875804
- [Derived] Rezvani K, Yong AS, Mielke S, Savani BN, Jafarpour B, Eniafe R, Le RQ, Musse L, Boss C, Childs R, John Barrett A. Lymphodepletion is permissive to the development of spontaneous T-cell responses to the self-antigen PR1 early after allogeneic stem cell transplantation and in patients with acute myeloid leukemia undergoing WT1 peptide vaccination following chemotherapy. Cancer Immunol Immunother. 2012 Jul;61(7):1125-36. doi: 10.1007/s00262-011-1187-z. Epub 2011 Dec 24. PMID 22198310
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/B_2007-H-0091.html

RESULTS

PARTICIPANT FLOW:
Groups:
- WT1 Peptide Vaccine: Subjects with hematologic malignancies will receive WT1 peptide vaccine to evaluate if the intervention will stimulate a protective immune response.
Period: Overall Study
Arm/Group | WT1 Peptide Vaccine
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | WT1 Peptide Vaccine
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Cellular Immune Response
Description: Minimum criterion for a cellular immune response was defined as the emergence of detectable T cell frequency against Willm's tumor 1 (WT1) when the pre-study analysis found no response, or a twofold increase in T cell frequency at any post vaccination time point
Time Frame: 7 weeks after last dose of vaccine
Measure: Number; unit: participants
Arm/Group | WT1 Peptide Vaccine
Number analyzed (Participants) | 4
participants | 4

2. Secondary Outcome: Disease Response
Description: Clinical response of underlying malignancy to the vaccination
Time Frame: 7 weeks after last dose of vaccine
Measure: Number; unit: participants
Groups:
- WT1 Peptide Vaccine: All 4 patients who were accrued went on to receive the vaccine.
  Complete Response (CR): defined as an absolute neutrophil count of ≥500/µL, platelet count of ≥75,000/µL, no leukemic blasts in the blood nor evidence of extramedullary leukemia, bone marrow (BM) with a cellularity of more than 20%, maturation of all three cell lineages, no Auer rods, and less than 5% bone marrow blast cells.
  Partial response (PR): 50% reduction in marrow blasts, with an absolute neutrophil count (ANC) greater than 500/µL, and platelet count greater than 75000/µL.
  No response: subjects who did not meet the above response criteria were defined as non-responders.
Arm/Group | WT1 Peptide Vaccine
Number analyzed (Participants) | 4
participants
  Complete response | 0
  Partial response | 1
  No response | 3

ADVERSE EVENTS:
Groups:
- WT1 Peptide Vaccine: All 4 patients who were accrued went on to receive the vaccine
Arm/Group | WT1 Peptide Vaccine
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
Although there was one partial response at 7 weeks, this patient went on to relapse as well.

Consequently, all 4 patients had rapid relapses despite vaccination. Accrual was stopped at 4.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No